CLINICAL TRIAL: NCT03129906
Title: Impact of the Restriction of Sources of Gluten in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Jacqueline Isaura Alvarez Leite, MD.Ph.D, Federal University of Minas Gerais
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 48529415.8.0000.5149
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; non-celiac gluten sensitivity
MeSH Terms: conditions — Fibromyalgia | interventions — Glutens

STUDY DESIGN:
Intervention Model Description: All participants received placebo capsules and, after that, gluten capsules.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten (Active Comparator): Capsules containing 8 g/day of gluten (6,3g of protein) were blindly administered for 7 days
  Interventions: Dietary Supplement: Gluten
- Rice protein (Placebo Comparator): Capsules containing 6,4 g/day of rice protein were blindly administered for 7 days
  Interventions: Dietary Supplement: Rice protein

INTERVENTIONS:
Dietary Supplement: Gluten
  Arms: Gluten
Dietary Supplement: Rice protein
  Arms: Rice protein

SUMMARY:
The aim of this study is to evaluate the impact of gluten-free diets on symptoms and inflammatory markers in individuals with previous diagnosis of fibromyalgia (FM), as well as to identify the presence of non-celiac gluten sensitivity (NCSG) in individuals with FM. Patients with FM diagnosis will be kept on a gluten-free diet for a 10 weeks. In the 7th week, they will receive placebo capsules for 7 days and after washout, capsules containing gluten for another 7 days. A questionnaire based on Salerno protocol will be applied to evaluate the presence of NCGS in the beginning, 8th week and 10 week.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic and widespread pain condition, usually accompanied by several associated symptoms such as fatigue, sleep disorder, headache, irritable bowel syndrome and mood disorders. Recent studies point to the possibility of gluten protein having a role in the development of FM symptoms in a subgroup of patients. Fourteen patients with FM diagnosis will be kept on a diet restrict in gluten-free foods for a period 10 weeks. At the 7th week they received rice protein isolate capsules (placebo) for 7 days, followed by a 3-day wash-out and a new challenge with capsules containing 8 g/day of gluten (corresponding to 6,3g gluten protein) for another 7 days. In the initial period, at 8th week (final of placebo period) and after challenge with gluten (10th week), blood will be collected for analysis of inflammatory markers. Questionnaires will be carried out to evaluate the quantity and severity of FM symptoms and the impact of FM on daily routine. Inflammatory markers (IL-1bera, IL-6 and IL-10) will be evaluated in the blood. In the challenger period (gluten or placebo) questionnaires will be carried out to evaluate the quantity and severity of symptoms related to fibromyalgia and the impact of fibromyalgia on a daily basis. In addition, a questionnaire based on Salerno protocol was applied to evaluate the presence of NCGS.

ELIGIBILITY:
Inclusion Criteria:

• Women between 18 and 65 years of age with prior clinical diagnosis of FM, according to the American College of Rheumatology criteria of 2010

Exclusion Criteria:

* Subjects diagnosed with positive serology for celiac disease or allergy to wheat
* Subjects diagnosed with autoimmune diseases
* Subjects with diseases that are not part of the comorbidities associated with FM and t hat could influence the results of the study
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-25; Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Changes in fibromyalgia Symptoms by Salerno protocol | Baseline, 4th and 8th weeks, 10th week
  Self report of symptoms intensity in the last week. Each item is scored 0 (no symptom) to 10 (very intense symptom).

SECONDARY OUTCOMES:
Changes in body weight | Baseline, 8th and 10th weeks
  measured in weight in kg
Height | baseline
  measured in meters
changes in BMI | Baseline, 8th and 10th weeks
  in kg of body weight/square of height
Changes in IL-6 blood concentration | Baseline, 8th and 10th weeks
  measure by ELISA in ug/mL
Changes in IL-10 blood concentration | Baseline, 8th and 10th weeks
  measure by ELISA in ug/mL
Changes in IL-1beta blood concentration | Baseline, 8th and 10th weeks
  measure by ELISA in ug/mL
changes in Food intake | Baseline, 8th and 10th weeks
  measured in % of kcal

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline I Alvarez-Leite, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Laboratório de Aterosclerose e Bioquimica Nutricional, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No